CLINICAL TRIAL: NCT03934333
Title: A Phase 1, Randomized, Open-label, Single-dose, 2-way Cross-over Study to Compare the Pharmacokinetics of Budesonide Delivered by PT027 Compared With Pulmicort Flexhaler (ELBRUS)
Brief Title: A Study to Compare the Pharmacokinetics of Budesonide Delivered by PT027 Compared With Pulmicort Flexhaler (ELBRUS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D6930C00011
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Relative Bioavailability
Keywords: Pharmacokinetics; Inhaled corticosteroid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A/B (BDA MDI/Pulmicort) (Experimental): For each participant, the BDA MDI/Pulmicort Flexhaler DPI will be administered as a single dose (2 inhalations) on Day 1 of the respective treatment period per the assigned treatment sequence. The IMP will be administered in the morning, at approximately the same time of day throughout the study (±30 minutes).
  Interventions: Drug: BDA MDI 160/180 mcg; Drug: Pulmicort Flexhaler 180 mcg
- B/A (Pulmicort/ BDA MDI) (Experimental): For each participant, the Pulmicort Flexhaler DPI / BDA MDI will be administered as a single dose (2 inhalations) on Day 1 of the respective treatment period per the assigned treatment sequence. The IMP should be administered in the morning, at approximately the same time of day throughout the study (±30 minutes).
  Interventions: Drug: BDA MDI 160/180 mcg; Drug: Pulmicort Flexhaler 180 mcg

INTERVENTIONS:
Drug: BDA MDI 160/180 mcg — Budesonide/albuterol sulfate pressurized inhalation suspension, single dose given as 2 inhalations of 80/90 mcg.
Drug: Pulmicort Flexhaler 180 mcg — Pulmicort Flexhaler aerosol, power, single-dose given as 2 inhalations of 90 mcg.

SUMMARY:
This study is to compare the systemic exposure of budesonide delivered by the combination inhaler (budesonide/albuterol sulfate pressurized inhalation suspension [BDA metered dose inhaler {BDA MDI}]) with Pulmicort Flexhaler dry-powder inhaler (DPI).

DETAILED DESCRIPTION:
This study will be an open-label, randomized, 2-way cross-over study in healthy adult male or female participants, performed at a single study center.Participants will receive single doses of BDA MDI or Pulmicort Flexhaler on 2 occasions, under fasted conditions. There will be a minimum washout period of 3 days between each dose administration. A total of 66 participants will be randomized in this study to ensure that at least 62 participants are evaluable. The study will comprise of screening period of maximum 27 days; Two treatment periods during which participants will be resident from the day prior to administration of budesonide/albuterol sulfate pressurized inhalation suspension metered dose inhaler (BDA MDI) or Pulmicort Flexhaler (Day -1) until at least 24 hours after dosing. Participants will be discharged on the morning of Day 2; and a final follow-up visit within 5 to 7 days after the last administration of BDA MDI or Pulmicort Flexhaler.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male and female participants aged 18 to 55 years with suitable veins for cannulation or repeated venipuncture.
3. Females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit, must not be lactating.
4. Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
5. Must be able to demonstrate proper inhalation technique using the Vitalograph Aerosol Inhalation Monitor (AIM) device 3 repeated times as well as be able to use the BDA MDI and Pulmicort Flexhaler devices according to instructions.
6. Forced expiratory volume in 1 second in liters (FEV1) ≥80% of predicted value and FEV1/forced vital capacity in liters (FVC) ratio ≥70%.

Exclusion Criteria:

1. Pregnant or nursing female participants or participants who are trying to conceive
2. For female participants, a positive serum human chorionic gonadotropin (hCG) test at the Screening Visit or a positive urine hCG at admission for any of the 2 Treatment Periods.
3. History of any clinically significant disease or disorder which, in the opinion of the PI, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
4. History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
5. Participants who have cancer that has not been in complete remission for at least 5 years.
6. Any history of asthma or Chronic obstructive pulmonary disease (COPD).
7. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
8. Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results at the Screening Visit, as judged by the PI.
9. Any clinically significant abnormal findings in vital signs at the Screening Visit, as judged by the PI.
10. Any clinically significant abnormalities on 12-lead electrocardiogram (ECG) at the Screening Visit, as judged by the PI.
11. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.
12. Known or suspected history of alcohol or drug abuse, or excessive intake of alcohol, in past 2 years, as judged by the PI.
13. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study. The period of exclusion begins 3 months after the final dose or one month after the last visit whichever is the longest.
14. Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to the Screening Visit.
15. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the PI or history of hypersensitivity to drugs with a similar chemical structure or class to budesonide, albuterol sulfate and any component of the MDI and DPI.
16. Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 3 months prior to screening.
17. Positive screen for drugs of abuse, cotinine or alcohol at the Screening Visit or on each admission to the Clinical Unit.
18. Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
19. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life.
20. Involvement of any AstraZeneca, PAREXEL or study site employee or their close relatives.
21. Judgment by the PI that the participant should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
22. Vulnerable participants, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve from time zero to infinity (AUC) for budesonide | On Day 1 (Pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose) and on Day 2 (24 hours post-dose)
  To compare the systemic exposure of budesonide after single-dose administration of BDA MDI versus Pulmicort Flexhaler
Area under the plasma concentration-curve from time zero to time of last quantifiable concentration [AUC(0-t)] for budesonide | On Day 1 (Pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose) and on Day 2 (24 hours post-dose)
  To compare the systemic exposure of budesonide after single-dose administration of BDA MDI versus Pulmicort Flexhaler
Maximum observed plasma concentration (Cmax) for budesonide | On Day 1 (Pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose) and on Day 2 (24 hours post-dose)
  To compare the systemic exposure of budesonide after single-dose administration of BDA MDI versus Pulmicort Flexhaler

SECONDARY OUTCOMES:
Time to reach maximum observed plasma concentration (tmax) | On Day 1 (Pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose) and on Day 2 (24 hours post-dose)
  To determine tmax for budesonide delivered by BDA MDI and Pulmicort Flexhaler
Time of last quantifiable plasma concentration (tlast) | On Day 1 (Pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose) and on Day 2 (24 hours post-dose)
  To determine tlast for budesonide delivered by BDA MDI and Pulmicort Flexhaler
Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t½λz) | On Day 1 (Pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose) and on Day 2 (24 hours post-dose)
  To determine t½λz for budesonide delivered by BDA MDI and Pulmicort Flexhaler
Terminal elimination rate constant (λz) | On Day 1 (Pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose) and on Day 2 (24 hours post-dose)
  To determine λz for budesonide delivered by BDA MDI and Pulmicort Flexhaler
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | On Day 1 (Pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose) and on Day 2 (24 hours post-dose)
  To determine CL/F for budesonide delivered by BDA MDI and Pulmicort Flexhaler
Apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) | On Day 1 (Pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose) and on Day 2 (24 hours post-dose)
  To determine Vz/F for budesonide delivered by BDA MDI and Pulmicort Flexhaler
Number of participants with adverse events and serious adverse events | From screening (Day -27 to Day -2) to post study visit ( 5-7 days)
  To assess the safety and tolerability of BDA MDI and Pulmicort Flexhaler

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ronald Goldwater, MD, Principal Investigator — MD
Locations (1):
- Research Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided